CLINICAL TRIAL: NCT01500057
Title: An Open-Label Randomized Phase 4 Study of Greenlight XPS Laser Versus BiVAP Saline Vaporization of the Prostate in Men With Symptomatic Benign Prostatic Hyperplasia
Brief Title: Phase 4 Study of Greenlight XPS Laser Versus BiVAP Saline Vaporization of the Prostate in Men With Symptomatic Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooklyn Urology Research Group (Other)
Collaborators: American Medical Systems (Industry); Richard Wolf Medical Instruments Corporation (RWMIC) (Unknown)
Responsible Party: Principal Investigator, Ivan Grunberger, MD, Medical Director, Brooklyn Urology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB Protocol# 20111638
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: enlarged prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Greenlight XPS Laser (Active Comparator): Greenlight XPS Laser of the prostate
  Interventions: Device: Greenlight XPS Laser
- BiVAP Saline Vaporization (Active Comparator): BiVAP Saline Vaporization of the prostate
  Interventions: Device: BiVAP Saline Vaporization of the prostate

INTERVENTIONS:
Device: Greenlight XPS Laser — Treatment of BPH with Greenlight XPS laser
  Arms: Greenlight XPS Laser
Device: BiVAP Saline Vaporization of the prostate — treatment of BPH with BiVAP Saline Vaporization
  Arms: BiVAP Saline Vaporization

SUMMARY:
This is a Phase 4, prospective, open-label, randomized study of Greenlight XPS Laser versus BiVAP Saline Vaporization of the prostate in men with symptomatic Benign Prostatic Hyperplasia (BPH). The study consists of a screening phase, treatment, followed by follow-up visits at 1 week, 4 weeks, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* male over the age of 18 years
* present with symptomatic/ obstructive symptoms secondary to PBH requiring surgical intervention
* subjects must read, understand and sign the Informed Consent
* AUA ≥ 15
* Qmax < 15mL/sec
* Stopped BPH medication. Alpha blockers 15 days 5-α-reductase 3 months
* Prostate volume ≥ 30g

Exclusion Criteria:

* PVR > 300ml
* Current urine retention
* Previous surgical or invasive treatments (TURP, TUMT, TUNA)
* PSA ≥ 4 (must have negative biopsy within last 12 months)
* Neurogenic bladder
* Obstruction due to urethral stricture
* Any disorder or condition of the subject that the investigator believes will counter indicate their inclusion in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-12; Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brooklyn Urology Research Group, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization
Started | 31 | 35
Completed | 25 | 31
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.1) | 65.5 (10.0) | 67.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 35 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in American Urological Association Symptom Score
Description: The American Urological Association Symptom Score range is 0-35 with 35 being the most severe urinary symptoms
Time Frame: Baseline and 12 months
Population: All people who completed the study and had data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization
Number analyzed (Participants) | 23 | 27
units on a scale | -14.7 (9.0) | -10.5 (8.6)

2. Primary Outcome: Change From Baseline to 12 Months in Maximum Urinary Flow Rate (Qmax)
Description: maximum urinary flow rate was measures using uroflow device
Time Frame: baseline and 12 months
Population: all participants who completed the study and have available data
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization
Number analyzed (Participants) | 23 | 24
ml/sec | 5.9 (8.6) | 2.3 (8.3)

3. Secondary Outcome: Change From Baseline to 12 Months in Post Void Residual Volume
Description: post void residual was measured using a bladder scan device
Time Frame: baseline and 12 months
Population: all participants who completed the study and have available data
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization
Number analyzed (Participants) | 23 | 24
ml | -61.9 (104.0) | -36.7 (122.2)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Greenlight XPS Laser | BiVAP Saline Vaporization
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35
Other Adverse Events (participants affected / at risk) | 2/31 | 4/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Greenlight XPS Laser (N=31) | BiVAP Saline Vaporization (N=35)
urethral stricture (Renal and urinary disorders) | 0 (0) | 3 (3)
urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes